CLINICAL TRIAL: NCT06783647
Title: An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of LBL-024 in Combination With Other Drugs for the Treatment of Patients With Advanced Solid Tumour[Substudy Number 01(NSCLC)]
Brief Title: A Clinical Trial of LBL-024 Combination Drug in Patients With Advanced Solid Tumours[Substudy 01(NSCLC)]
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN004_01(NSCLC)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumour
MeSH Terms: interventions — Injections; Docetaxel; Bevacizumab; Pemetrexed; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LBL-024+Docetaxel/LBL-024+Bevacizumab+Docetaxel (Experimental): Cohort 1 A：
  Subjects were treated with LBL-024 combined with docetaxel
  or LBL-024 combined with bevacizumab and docetaxel,
  Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Docetaxel Injection; Drug: Bevacizumab Injection
- LBL-024+Docetaxel (Experimental): Cohort 1 B：
  Subjects were treated with LBL-024 combined with docetaxel,
  Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Docetaxel Injection
- LBL-024+Pemetrexed Disodium+Carboplatin/LBL-024+pemetrexed Disodium (Experimental): Cohort 2 A：
  Subjects were treated with LBL-024 combined with pemetrexed and carboplatin,
  after a period of time,LBL-024 and pemetrexed were used for maintenance treatment.
  Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Pemetrexed Disodium for Injection; Drug: Carboplatin Injection
- LBL-024+Paclitaxel+Carboplatin/LBL-024 (Experimental): Cohort 2 B：
  Subjects were treated with LBL-024 combined with paclitaxel and carboplatin,
  after a period of time,LBL-024 was used for maintenance treatment.
  Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Paclitaxel Injection; Drug: Carboplatin Injection

INTERVENTIONS:
Drug: LBL-024 for Injection — intravenous infusion.
  Other Names: LBL-024
Drug: Docetaxel Injection — intravenous infusion.
  Other Names: Docetaxel
  Arms: LBL-024+Docetaxel; LBL-024+Docetaxel/LBL-024+Bevacizumab+Docetaxel
Drug: Bevacizumab Injection — intravenous infusion.
  Other Names: Bevacizumab
  Arms: LBL-024+Docetaxel/LBL-024+Bevacizumab+Docetaxel
Drug: Pemetrexed Disodium for Injection — intravenous infusion.
  Other Names: Pemetrexed Disodium
  Arms: LBL-024+Pemetrexed Disodium+Carboplatin/LBL-024+pemetrexed Disodium
Drug: Paclitaxel Injection — intravenous infusion.
  Other Names: Paclitaxel
  Arms: LBL-024+Paclitaxel+Carboplatin/LBL-024
Drug: Carboplatin Injection — intravenous infusion.
  Other Names: Carboplatin
  Arms: LBL-024+Paclitaxel+Carboplatin/LBL-024; LBL-024+Pemetrexed Disodium+Carboplatin/LBL-024+pemetrexed Disodium

SUMMARY:
An open-label, multicenter, phase II clinical study to evaluate the efficacy and safety of LBL-024 in combination with other drugs for the treatment of patients with advanced solid tumour.

DETAILED DESCRIPTION:
This trial is an open-label, multicenter, phase II clinical study of LBL-024 combination therapy in patients with advanced NSCLC, to evaluate the efficacy and safety of LBL-024 combination therapy .The trial includes 4 cohorts.

Cohort 1 A:This cohort will have a safety run-in period in which a small number of subjects will be enrolled to receive LBL-024 Combination Administration. After the subjects completed the 21-day safety observation, the sponsor and investigator jointly assessed the safety and tolerability of the combination drugs. If the safety and tolerability of combination drugs are good, the Cohort will continue to enroll subjects for the extension study of combination administration. Eligible subjects will be randomized in a 1: 1 ratio to Arm A or Arm B.

Cohort 1 B:This cohort will have a safety run-in period, a small number of subjects will be enrolled to receive LBL-024 Combination Administration.After the subjects completed the 21-day safety observation, the sponsor and investigator jointly assessed the safety and tolerability of the combination drugs.If the safety and tolerability of combination drugs are good, the Cohort will continue to enroll subjects for the extension study of combination administration.

Cohort 2 A:This cohort will have a safety run-in period, a small number of subjects will be enrolled to receive LBL-024 Combination Administration, and after a period of time, LBL-024 and pemetrexed will be used for maintenance treatment.After completing the 21-day safety observation, the safety and tolerability of combination drugs will be assessed. If the safety and tolerability of combination drugs are good, this cohort will continue to enroll subjects.

Cohort 2 B: This cohort will have a safety run-in period, a small number of subjects will be enrolled to receive LBL-024 Combination Administration and after a period of time, and then use LBL-024 for maintenance treatment. After completing the 21-day safety observation, the safety and tolerability of combination drugs will be assessed. If the safety and tolerability of combination drugs are good, this cohort will continue to enroll subjects.

This study will enroll up to 230 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen, visit schedule, laboratory test, and other requirements of the protocol, and voluntarily enroll in the study and sign the written informed consent.
2. Age 18-75 years (inclusive of boundaries) at the time of signing informed consent form.
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1.
4. The expected survival time is at least 12 weeks.
5. According to the evaluation of RECIST 1.1 standard, the subjects enrolled have at least one measurable lesion.
6. There is adequate organ and bone marrow function,Conforms to laboratory test results.
7. Males with fertility and females of childbearing age are willing to take effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug (including abstinence, intrauterine device, various hormonal contraception, correct use of contraception Sets，etc）; Women of childbearing age include pre-menopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.

Exclusion Criteria:

1. Participation in clinical studies of antineoplastic agents within 4 weeks before the first use of study drug,or Subject is expected to receive any other form of systemic or local anti-tumor therapy outside the protocol during the study.
2. Use of immunomodulatory drugs within 2 weeks before the first use of study drug,Including but not limited to thymopeptide, interleukins, interferon, etc.
3. Patients with active infection.
4. Patients with clinically uncontrollable pleural effusion, pericardial effusion, ascites, and those requiring repeated drainage or medical intervention.
5. The patient has a Medical history of immunodeficiency, including HIV antibody positive.
6. Active hepatitis B or active hepatitis C.
7. Women during pregnancy or lactation.
8. History of mental illness (interfering with understanding or giving informed consent), drug abuse, alcoholism or drug addiction.
9. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Objective Response Rate (complete response (CR) + partial response (PR)), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1), refers to the percentage of study subjects who achieve a complete response or partial response.

SECONDARY OUTCOMES:
Disease Control Rate(DCR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Percentage of participants achieving CR and PR and stable disease (SD).
Duration of Response(DOR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The period from the participants first achieving CR or PR to disease progression.
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum drug concentration in plasma after administration
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  After administration,Time to reach maximum drug concentration in plasma
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.

CONTACTS AND LOCATIONS:
Overall Officials: li Zhang, Principal Investigator — Sun Yat-sen University
Locations (24):
- China (24):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No